CLINICAL TRIAL: NCT06887985
Title: An Early Exploratory Clinical Study of the Safety, Tolerability, and Initial Efficacy of JY231 Injection for the Treatment of Refractory Autoimmune Diseases (ADs)
Brief Title: JY231(JY231) Injection for the Treatment of Refractory Autoimmune Diseases (ADs)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: He Huang (Other)
Responsible Party: Sponsor-Investigator, He Huang, Professor, Director of the Bone Marrow Transplantation Center, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-24-007
Record Dates: First submitted 2025-03-19; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single-center, open, single arm study (Experimental): JY231 injection for the treatment of refractory autoimmune diseases (ADs) subjects who meet the inclusion criteria will receive a single intravenous injection of JY231, followed by regular observation and follow-up of the subject.
  Interventions: Drug: JY231 Injection

INTERVENTIONS:
Drug: JY231 Injection — This is an open-label, single-arm study to evaluate the efficacy and safety of in vivo chimeric antigen receptor T-Cell (CAR-T cell) therapy in patients with relapsed refractory B-cell leukemia.
  Upon enrollment, subjects will receive an intravenous infusion of the JY231 preparation. Following the infusion, subjects will be hospitalized for one month for observation, and subjects will be evaluated for safety and efficacy. Subjects will be followed for up to 15 years to determine if the disease is under control.

SUMMARY:
This study is an investigator-initiated single center, single arm clinical study with a target population of patients with Refractory Autoimmune Diseases (ADs). It is an early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of Refractory Autoimmune Diseases (ADs).

DETAILED DESCRIPTION:
This study included the screening period (Day -18 to Day -7), the baseline period (Day -1), the treatment and observation period (Day 0 to 28), and the follow-up period (Month 2[from Day 29] to Year 15). Participants eligible for the screening period will be admitted to the study center for a single JY231 treatment and a follow-up period after the end of the treatment and observation period. After completing the follow-up for the first five years, methods such as telephone or written questionnaires can be used, and relevant samples should be collected as much as possible. The subjects should be followed up at least once a year until the end of the follow-up period. The maximum monitoring time can be extended to 15 years, and all monitoring data during the extension process need to be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18~75 years old, male or female, signed informed consent (ICF);
2. Diagnosis of one of the following diseases:

   1. Systemic Lupus Erythematosus (SLE), European League Against Rheumatism/ (EULAR)/American College of Rheumatology(ACR) 2019 criteria), and Antinuclear Antibodies(ANA) > 1:80 or ds-DNA positive;
   2. Dry syndrome (SS), 2016 ACR/EULAR criteria and at least Sjögren's Syndrome Antigen A(SSA) positive;
   3. Systemic sclerosis (SSc), 2013 ACR/EULAR criteria and ANA > 1:80 or anti-Scleroderma(SCL)-70 positive;
   4. Dermatomyositis (DM), 2017 EULAR/ACR classification criteria and positive for any of the myositis-specific antibodies (Jo-1), Zo, Anti-Glycyl-Transfer Ribonucleic Acid(tRNA) Synthetase Antibody(EJ), Anti - Threonyl - tRNA Synthetase Antibody(PL-7), Anti-Aspartyl-tRNA Synthetase Antibody(KS), Anti-isoleucyl-tRNA Synthetase Antibody(OJ), PL-12, Anti-Tyrosyl-tRNA Synthetase Antibody(YRS), Anti-nuclear matrix protein(NXP)-2, Anti - transcription intermediary factor 1 gamma Antibody(Anti-TIF1g), Anti-Mi-2, Anti-small ubiquitin - like modifier - activating enzyme Antibody(Anti-SAE), Anti-MDA-5, Anti-signal recognition particle Antibody(Anti-SRP), Anti-HMGCR);
   5. Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis (ANCA-AAV), including granulomatous polyangiitis (GPA), or microscopic vasculitis (MPA), or eosinophilic granulomatous polyangiitis (EGPA),2022 ACR/EULAR criteria, and ANCA antibody-positive, including c-ANCA/p-ANCA/anti Proteinase 3(PR3)/anti-Myeloperoxidase(MPO) positive.
3. Patients who have been treated with ≥2 immunosuppressive agents for 6 months, or who are intolerant to standard therapy, or who have relative contraindications, and whose disease activity meets the following criteria:

   1. For SLE patients, SLEDAI≥ 8 points;
   2. For SS patients, European League Against Rheumatism Sjögren's Syndrome Disease Activity Index(ESSDAI) ≥ 14 points;
   3. For SSc patients with an Modified Rodnan Skin Score(mRSS) score between 10-35 (inclusive of the cutoff), combined with interstitial lung disease (ILD);
   4. For DM patients, 1 year after diagnosis, and the following conditions are met:

      ① Rash VAS score (based on MDAAT) ≥ 3 cm and at least 3 CSM abnormalities;

      ②Muscle biopsy pathology or muscle nuclear magnetic resonance suggestive of active inflammation;

      ③ Bilateral Manual Muscle Testing (MMT-8) < 125/150 and at least 2 additional Core set measures (CSM) meeting the criteria specified below: a. Patient scores on a 10 cm Visual Analog Scale (VAS) with a minimum of 2.0 cm; b. Physician scores on a 10 cm VAS with a minimum of 2.0 cm; c. Health Assessment Questionnaire (HAQ) Disability Index with a minimum value of 0.25; d. Elevation of at least one muscle enzyme (including creatine kinase (CK), aldolase, lactate dehydrogenase (LDH), alanine aminotransferase (ALT), and aspartate aminotransferase (AST)), with a minimum level of 1.3 x the upper limit of normal; and e. Extramuscular Organ Disease Activity Score with a minimum level of 1.3 x the upper limit of normal on a 10 cm VAS scale. minimum of 1.0 cm on a 10 cm VAS scale (This VAS is a physician's comprehensive assessment based on the Myositis Disease Activity Assessment Tool (MDAAT) which evaluates activity scores on the General Condition, Skin, Skeletal, Gastrointestinal, Lung, and Cardiac scales);
   5. For ANCA-AAV patients, British Vasculitis Activity Score(BVAS) score ≥15,and ANCA antibody.
4. Eastern Cooperative Oncology Group (ECOG) 0 to 1 point;
5. Critical organ function assessment meets the following conditions:

   1. Blood: hemoglobin ≥60g/L, platelet count ≥20×109/L;
   2. Cardiac function: left ventricular ejection fraction (LVEF) ≥55%, ECG without obvious abnormalities;
   3. Renal function: Estimated Glomerular Filtration Rate(eGFR) ≥30 mL/min/1.73m2;
   4. Liver function: AST and ALT ≤ 3.0 upper limit of normal(ULN) and total bilirubin ≤ 2.0 ULN;
   5. Have criteria for single or venous blood collection and no other contraindications to cell collection;
6. Subjects of childbearing age with negative urine pregnancy test results and agree to use effective contraception during the study until 1 year post-infusion;
7. The patient or his/her guardian agrees to participate in the study and signs an informed consent form, indicating that he/she understands the purpose and procedures of the study and is willing to participate in the study.

Exclusion Criteria:

1. Have received prior CAR-T cell therapy;
2. Suffering from severe cardiac, hepatic, pulmonary, hematologic, or endocrine system disorders that, in the judgment of the investigator, outweigh the risks of participation in the study;
3. Active or uncontrollable infection requiring systemic therapy within 1 week prior to screening;
4. Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) positive and peripheral blood Hepatitis B virus (HBV) DNA titer test is greater than the normal reference range; or Hepatitis C virus (HCV) antibody positive and peripheral blood Hepatitis C virus (HCV) RNA titer test is greater than the normal reference range; or Human Immunodeficiency Virus (HIV) antibody positive; or positive syphilis test; or positive cytomegalovirus (CMV) DNA test;
5. Have received a live vaccine within 4 weeks prior to screening;
6. Women who are pregnant or breastfeeding, and female subjects who plan to become pregnant within 2 years of their JY231 injection infusion or male subjects whose partners plan to become pregnant within 2 years of their JY231 injection infusion;
7. Patients with malignant diseases such as malignant tumors prior to screening, except adequately treated cervical carcinoma in situ, basal cell or squamous epithelial cell skin cancer, localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
8. Patients who have participated in another clinical study within 3 months prior to screening;
9. Other conditions that the investigator considers unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.
Maximal Tolerated Dose(MTD) | Up to 28 days after infusion
  MTD will be determined based on Dose-Limiting Toxicity(DLTs) observed during the first 28 days of study treatment.